CLINICAL TRIAL: NCT06675162
Title: The Physiological Responses of Muscle Strengthening Training with Pilates Reformer in Overweight-obese Women and Women with Normal Body Weight
Brief Title: Effect of Muscle Strengthening Training with Pilates Reformer on Overweight/obese and Normal Body Weight Women (PRET)
Acronym: PRET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Syrou Niki, RN,MPH, PhD, Principal Investigator, University of Thessaly
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2432/09.10.2024
Record Dates: First submitted 2024-10-31; First posted 2024-11-05 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Physiological Responses; Pilates Exercise; Overweight and Obese Women; Energy Expenditure; Strength Training
Keywords: Pilates Reformer Training; Energy Expenditure; Oxygen consumption; Blood lactate; Overweight; Obesity; Body composition
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pilates Reformer Training (OW) (Experimental): A group of women with overweight/obesity in this arm will participate in a 60-minute muscle-strengthening training session with Pilates Reformer equipment.
  Interventions: Other: Pilates Reformer Training
- Pilates Reformer Training (NW) (Experimental): A group of women with normal weight in this arm will participate in a 60-minute muscle-strengthening training session with Pilates Reformer equipment.
  Interventions: Other: Pilates Reformer Training

INTERVENTIONS:
Other: Pilates Reformer Training — Participants will perform a 60-minute Pilates Reformer muscle-strengthening session. The training will include a 7-10 minute warm-up, 35 minutes of muscle strengthening and mobility exercises and a 5-minute recovery. During the training, the physiological responses and the energy expenditure of the participants will be recorded.

SUMMARY:
This study investigates the physiological responses and the metabolic burden of a Pilates Reformer strength training session in physically inactive premenopausal women with a body mass index of 18-24.9 and 25.01-39.9. The sample included 20 women divided into two groups: 10 with normal weight (NW) and 10 with overweight/obesity (OB). In a non-randomised control design, the participants will perform a 60-minute muscle-strengthening session with Pilates Reformer equipment.

DETAILED DESCRIPTION:
Pilates Reformer (PR) is one of the most popular types of exercise worldwide and is considered a gentle and safe method for untrained and overweight people. The PR training approach has been found to contribute positively to various health conditions (vascular function, blood pressure, physical fitness, musculoskeletal problems), improving the quality of life and mental well-being of the participants. At the same time, it seems that it can have a positive effect on the lipid profile and other biochemical markers such as insulin and fasting glucose. Furthermore, muscle strengthening training with PR equipment provides better levels of mobility, increasing active range of motion, and also provides greater pelvic and trunk stability for both adult and middle-aged participants.

This study is designed to investigate the physiological and metabolic burden of a muscle-strengthening session with PR equipment in 20 pre-menopausal and physically inactive women with a body mass index (BMI) of 18-24, 99 & 25.01-39.9, as well as to determine the contribution of energy systems (mitochondrial, glycolytic) during and after the exercise. Each training session will last approximately 60 minutes, will be led by at least one trainer, and will include a warm-up of 7-10 minutes, muscle strengthening and mobility exercises of 35 minutes, and a recovery of 5 minutes. Anthropometric indicators, dietary intake, resting heart rate, blood lactate, resting metabolic rate, muscle soreness, rate of perceived exertion, blood pressure, and performance measurements will be measured at baseline. The metabolic cost during PR training session will be estimated from heart rate, blood lactate, resting oxygen uptake, exercise oxygen uptake, and excess post-exercise oxygen consumption measurements using a portable gas analyzer. After the PR training session will be measured the rate of perceived exertion, blood pressure, blood lactate, and muscle soreness levels.

ELIGIBILITY:
Inclusion Criteria:

* Be approved for participation by an orthopedist and internist
* Have not followed any diet or nutritional supplements for weight loss in the last six months before the study
* The group with overweight/obesity will consist of women with a body mass index of 25.01 - 39.9 kg/m2
* Be physically Inactive in the last six months before the study.

Exclusion Criteria:

* Musculoskeletal injury
* Weight loss>10% in 6 months
* <20 years
* >50 years
* Μenopause
* Chronic diseases
* Use of alcohol, caffeine and any type of ergogenic supplements or medication during the study
* Physically active.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Change in exercise-induced energy expenditure | At pre-exercise, 60 minutes during PR training, and 30 minutes after the exercise session (single bout lasting 60 minutes)
  Exercise energy expenditure (kcal) will be measured using a portable indirect calorimetry system
Change in excess post-exercise oxygen consumption (EPOC) | At 30 minutes after the exercise session (single bout lasting 60 minutes)
  EPOC (kcal) will be measured using a portable indirect calorimetry system
Change in blood lactate concentration (BLa) | At pre- and post-exercise session (single bout) at 4 minutes post-exercise
  BLa (mmol/L) concentration will be measured in a microphotometer with commercially available kits
Change in heart rate | At pre-exercise, 60 minutes during PR training, and 30 minutes after the exercise session (single bout lasting 60 minutes)
  Heart rate (bpm) will be measured with a wearable heart rate monitor
Change in perceived exertion | At pre- and post-exercise session (single bout) at 4 minutes post-exercise.
  Rating of perceived exertion (RPE) will be measured with the Borg scale (0-10)
Respiratory Exchange Ratio (RER) | At pre-exercise, 60 minutes during PR training, and 30 minutes after the exercise session (single bout lasting 60 minutes)
  Respiratory Exchange Ratio (RER) will be measured using a portable indirect calorimetry system
Breath Frequency (BF) | At pre-exercise, 60 minutes during PR training, and 30 minutes after the exercise session (single bout lasting 60 minutes)
  Breath Frequency (BF) will be measured using a portable indirect calorimetry system
Change in oxygen consumption | At pre-exercise, 60 minutes during PR training, and 30 minutes after the exercise session (single bout lasting 60 minutes)
  Oxygen consumption will be measured using a portable indirect calorimetry system

SECONDARY OUTCOMES:
Body weight | At baseline and at 40 minutes after the exercise session.
  Body weight will be measured on a beam balance with a stadiometer
Body height | At baseline
  Body height will be measured on a beam balance with a stadiometer
Body mass index (BMI) | At baseline
  BMI will be calculated using the Quetelet's equation
Waist circumference (WC) | At baseline
  WC (cm) will be measured using a Gullick II tape
Hip circumference (HC) | At baseline
  HC (cm) will be measured using a Gullick II tape
Waist-to-hip ratio (WHR) | At baseline
  WHR will be calculated by dividing the waist by the hip measurement
Resting metabolic rate (RMR) | At baseline
  RMR (kcal) will be measured using a portable open-circuit indirect calorimeter with a ventilated hood system
Body fat (BF) | At baseline
  Body fat (%) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Fat mass (FM) | At baseline
  FM (kg) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Fat-free mass (FFM) | At baseline
  FFM (kg) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Bone mass density | At baseline
  Bone mass density will be measured by using Dual-emission X-ray absorptiometry
Bone mass content | At baseline
  Bone mass content will be measured by using Dual-emission X-ray absorptiometry
Peak Maximal oxygen consumption (Peak VO2) | At baseline
  Peak VO2 will be estimated by open circuit spirometry via breath by breath method
Dietary intake | At baseline
  Dietary intake will be assesed over a 7-day period using diet recalls
Systolic Blood Pressure | At pre-exercise, 60 minutes during PR training, and 30 minutes after the exercise session (single bout lasting 60 minutes)
  Systolic Blood Pressure will be examined using a sphygmomanometer
Diastolic Blood Pressure | At pre-exercise, 60 minutes during PR training, and 30 minutes after the exercise session (single bout lasting 60 minutes)
  Diastolic Blood Pressure will be examined using a sphygmomanometer
Rest Heart Rate | At baseline
  The rest heart rate will be estimated using a heart rate monitor
Evaluation of physical activity (PA) | At baseline
  The PA will be evaluated for seven days before the intervention via accelerometry

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Department of Physical Education and Sport Science, Trikala, Thessaly
  - Department of Physical Education and Sports Science, University of Thessaly, Trikala, Thessaly

IPD SHARING:
Plan to Share IPD: Undecided